CLINICAL TRIAL: NCT06357910
Title: A Randomized, Open Label, Single Dose, Crossover Clinical Trial to Evaluate the Pharmacokinetic Characteristics and Safety After Administration of a Fixed-dose Combination Drug of HCP2303 and Co-administration of RLD2302 and RLD2102 in Healthy Volunteers Under Fed Conditions
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety Between HCP2303 and Co-administration of Each Component in Healthy Volunteers Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-EMMA-102
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): * Period1 : RLD2302 + RLD2102
  * Period2 : HCP2303
  Interventions: Drug: HCP2303; Drug: RLD2302; Drug: RLD2102
- Arm 2 (Experimental): * Period1 : HCP2303
  * Period2 : RLD2302 + RLD2102
  Interventions: Drug: HCP2303; Drug: RLD2302; Drug: RLD2102

INTERVENTIONS:
Drug: HCP2303 — Take 1 tablet once per period
Drug: RLD2302 — Take 1 tablet once per period
Drug: RLD2102 — Take 1 tablet once per period

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic characteristics and safety between HCP2303 and co-administration of each component in fed condition in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 19~54 years in healthy volunteers
* 18.5 kg/m^2 ≤ BMI < 30 kg/m^2, weight(men) ≥55kg / weight(women) ≥45kg
* 90 mmHg ≤ sitSBP <140 mmHg, 50 mmHg ≤ sitDBP <90 mmHg
* Agrees that the person, spouse, or partner uses appropriate medically recognized contraception and does not provide sperm or eggs from the date of administration of the first investigational drug to 7 days after the administration of the last investigational drug
* Subjects who voluntarily decides to participate in this clinical trial and agree in writing to ensure compliance with the clinical trial

Exclusion Criteria:

* Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
* Subjects who cannot consume the high-fat meal provided during this clinical trial
* Subjects who judged ineligible by the investigator

Ages: 19 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
AUCt | 0~48 hours
  Pharmacokinetic evaluation
Cmax | 0~48 hours
  Pharmacokinetic evaluation

SECONDARY OUTCOMES:
AUCinf | 0~48 hours
  Pharmacokinetic evaluation
Tmax | 0~48 hours
  Pharmacokinetic evaluation
t1/2 | 0~48 hours
  Pharmacokinetic evaluation
CL/F | 0~48 hours
  Pharmacokinetic evaluation
Vd/F | 0~48 hours
  Pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Min-gul Kim, MD, Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Jeonbuk University Hospital, Jeonju, Jeollabuk-do, South Korea